CLINICAL TRIAL: NCT01921218
Title: Belatacept Therapy for the Failing Renal Allograft
Acronym: IM103-133
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Andrew B Adams (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Andrew B Adams, Assistant Professor of Surgery, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00060470; IM103-133 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2013-08-09; First posted 2013-08-13 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Failing Renal Allograft
Keywords: Kidney transplant
MeSH Terms: interventions — Abatacept; Tacrolimus; Cyclosporine; Mycophenolic Acid; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Belatacept (Nulojix) IV
  Interventions: Drug: Belatacept; Drug: Mycophenolate mofetil; Drug: prednisone
- Control (Active Comparator): Calcineurin inhibitor based therapy (cyclosporine or tacrolimus)
  Interventions: Drug: Calcineurin inhibitor therapy; Drug: Mycophenolate mofetil; Drug: prednisone

INTERVENTIONS:
Drug: Belatacept — Belatacept, dosing 10mg/kg- day 0, 2 weeks, 1 month, 2 months, 3 months; subsequent doses 5mg/kg monthly through duration of trial or until retransplantation, whichever is first.
  Other Names: Nulojix
  Arms: Treatment
Drug: Calcineurin inhibitor therapy — Upon enrollment, wean calcineurin inhibitor (CNI) to target tacrolimus trough of 3-5 nanogram/milliliter (ng/ml)or equivalent cyclosporine trough. Upon initiation of hemodialysis, discontinue CNI therapy over 5 days.
  Other Names: tacrolimus; cyclosporine
  Arms: Control
Drug: Mycophenolate mofetil — Continue current dose at enrollment. Upon initiation of dialysis, decrease dose by half, then discontinue 2 weeks later
  Other Names: Cellcept
Drug: prednisone — Begin steroid withdrawal one month after initiation of dialysis, with monthly reduction in dose by half, with plans to discontinue prednisone by 3 months after initiation of dialysis
  Other Names: Deltasone

SUMMARY:
The purpose of this study is to test the safety and effectiveness of belatacept (Nulojix®) in preventing antibody formation in patients with chronic failing kidney transplants. This study is a randomized study of first-time kidney transplant patients who have worsening kidney function and biopsy proven grade 2 or 3 interstitial fibrosis/tubular atrophy (IF/TA). Patients must be eligible to get a second transplant. They must have completed or be actively undergoing evaluation for re-listing for a second transplant. Patients will be randomized to either convert to belatacept or continue on calcineurin inhibitor-based therapy.

DETAILED DESCRIPTION:
The purpose of this study is to test the safety and effectiveness of the medicine belatacept (Nulojix®) in preventing antibodies from forming in people with a failing kidney transplant. Kidney transplant patients take immunosuppression medicines to prevent kidney rejection. When a kidney transplant begins to fail, the immunosuppression medicines are slowly weaned. Once dialysis is started, the immunosuppressant medicines are usually stopped. After immunosuppression is stopped, some people form antibodies. Antibodies are proteins that the immune system makes to protect against harmful foreign substances like bacteria, viruses, or foreign tissues, like a transplant. High levels of antibodies can make it harder to find a kidney donor for that person.

Participants will be randomized into one of the two treatment groups. One group will continue taking their current immunosuppression medicines. The people in the treatment group will be switched to belatacept (Nulojix®). Belatacept (Nulojix®) is an immunosuppression medicine that is approved by the U.S. Food and Drug Administration (the FDA) to prevent rejection in kidney transplant. Participants will stop taking calcineurin inhibitors (either cyclosporine or tacrolimus) or sirolimus but will keep taking other immunosuppression medicines like Cellcept (MMF) or azathioprine (Imuran) and prednisone. These medicines will be slowly weaned and will be stopped if the participant has to start dialysis. Participants will continue taking belatacept (Nulojix®), even while on dialysis.

The study team will test both groups to see how many people in each group develop antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Kidney transplant recipient (human leukocyte antigen (HLA) non-identical donor) who now has impaired renal allograft function with:
* Estimated glomerular filtration rate (GFR) < 35 with a decline in GFR of > 10% in the 12 months prior to enrollment and must have biopsy proven grade II or III interstitial fibrosis/tubular atrophy (IF/TA) OR
* Estimated GFR persistently < 20 ml/min over the 6 month period prior to enrollment absent other causes for graft dysfunction, and deemed to have a failing allograft by the patient's transplant nephrologist
* On a maintenance immunosuppressive regimen that includes calcineurin inhibitor (CNI)(tacrolimus or cyclosporine) or sirolimus and at least
* MMF of a dose of at least 1 gm/day or comparable dose of azathioprine OR
* Prednisone at a dose of at least 5 mg/day
* Men and women, ages 18 to 70, inclusive

Exclusion Criteria:

* Women of childbearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 8 weeks after the last dose of study drug.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test.
* Sexually active fertile men not using effective birth control if their partners are WOCBP.
* Subjects who are Epstein-Barr Virus (EBV) seronegative.
* Subjects with any prior solid organ (e.g., heart, liver, pancreas) or cell (e.g., islet, bone marrow) transplant other than a renal allograft. Exception may be made for recipient of a simultaneous kidney-pancreas transplant who had previously experienced graft loss of the pancreas allograft due to thrombosis or rejection.
* Subjects with presence of donor specific antibody at the time of enrollment
* Subjects who have a recent history (within 1 yr) of biopsy proven acute rejection > Banff grade Ia
* Subjects who have a living donor identified for re-transplant within 3 months
* Subjects with a history of post-transplant lymphoproliferative disease (PTLD)
* Subjects at risk for tuberculosis (TB)
* Subjects with a history of cancer within the past 3 years, other than non-melanoma skin cancer(s)
* Subjects with a positive BK virus serum polymerase chain reaction (PCR) > 20,000 copies at the time of enrollment OR history of biopsy-proven BK nephropathy within the year prior to enrollment.
* Subjects with a mammogram that is suspicious for malignancy and in whom the possibility of malignancy cannot be reasonably excluded following additional clinical, laboratory, or other diagnostic evaluations
* Subjects who have difficult intravenous access or other reasons that would likely preclude the ability to receive long-term intravenous infusions
* Hypersensitivity to any medications that will be used in the protocol
* Subjects who have used any investigational drug within the 30 days prior to anticipated enrollment
* Subjects currently receiving belatacept as part of their maintenance immunosuppressive regimen
* Prisoners, or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-08; Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B Adams, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Emory University Hospital and the Emory Clinic in Atlanta, Georgia. Enrollment began August 2013 and all follow up was complete by December 12, 2019.
Groups:
- Belatacept Treatment Group: Participants with a failing kidney or failed kidney transplant receiving belatacept therapy
- Control Group: Participants with a failing kidney transplant continuing their current immunosuppression and once allograft failed discontinuing immunosuppression
Period: Overall Study
Arm/Group | Belatacept Treatment Group | Control Group
Started | 6 | 7
Completed | 3 | 3
Not Completed | 3 | 4
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Kidney transplant | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belatacept Treatment Group | Control Group | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.12 (9.12) | 45.69 (14.99) | 51.31 (12.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 5 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Donor-specific Antibody Formation
Description: The number of participants in each group with donor-specific antibody formation at 36 months following randomization.
Time Frame: Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept Treatment Group | Control Group
Number analyzed (Participants) | 4 | 4
Participants | 3 | 4

2. Secondary Outcome: Glomerular Filtration Rate (GFR)
Description: The glomerular filtration rate (GFR) assesses kidney function. GFR uses values for serum creatinine (SCr) measured in mg/dL, age in years, blood urea nitrogen (BUN) measures in mg/dL, and serum albumin (Alb) measured in g/dL. GFR is calculated as 170 x (SCr/0.95)^(-0.999) x (Age)^(-0.176) x (0.762 if the patient is female) x (1.180 if the patient is black) x (BUN)^(-0.170) x (Alb)^(0.318). A value of 90 or above is considered normal while values between 15 and 29 indicate severely decreased kidney function and values below 15 indicate kidney failure. The GFR in participants who do not require dialysis will be followed for two years.
Time Frame: Baseline up to Month 24
Population: Participants requiring dialysis, either at the time of enrollment or initiating dialysis during the study, are not included in this analysis.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Belatacept Treatment Group | Control Group
Number analyzed (Participants) | 4 | 2
mL/min/1.73 m^2
  Baseline | 14.25 (7.80) | 14.5 (0.71)
  Month 1 | 14.25 (8.06) | 11 (1.41)
  Month 2: number analyzed (Participants) | 3 | 2
  Month 2 | 19.33 (4.93) | 10.5 (4.95)
  Month 3: number analyzed (Participants) | 3 | 2
  Month 3 | 16.33 (1.53) | 16.5 (4.95)
  Month 6: number analyzed (Participants) | 3 | 2
  Month 6 | 14.67 (1.15) | 14.5 (6.36)
  Month 9: number analyzed (Participants) | 3 | 2
  Month 9 | 14.67 (3.06) | 13.5 (10.61)
  Month 12: number analyzed (Participants) | 3 | 1
  Month 12 | 13.67 (2.89) | 20 (0)
  Month 18: number analyzed (Participants) | 1 | 0
  Month 18 | 7 (0) |
  Month 24: number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Initiation of Dialysis
Description: Time to dialysis is measured as the time of randomization to initiation of dialysis. Participants already requiring dialysis at the time of enrollment were excluded from this endpoint analysis.
Time Frame: Up to Year 2
Population: This analysis includes participants who initiated dialysis during the course of the study.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Belatacept Treatment Group | Control Group
Number analyzed (Participants) | 4 | 2
months | 11.75 (7.46) | 10.5 (2.12)

4. Secondary Outcome: Number of Participants With Anti-human Leukocyte Antigen (HLA) Alloantibodies
Description: The presence of anti-HLA Class I and Class II alloantibodies is categorized as being negative (absent for both classes of alloantibodies), positive for Class I, positive for Class II, and positive for both Class I and Class II alloantibodies.
Time Frame: Baseline up to Month 36
Population: This analysis includes participants remaining in the study at the indicated study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept Treatment Group | Control Group
Number analyzed (Participants) | 6 | 7
Participants
  Baseline - Negative | 6 | 5
  Baseline - Positive Class I | 0 | 2
  Baseline - Positive Class II | 0 | 0
  Baseline - Positive Class I and II | 0 | 0
  Month 12 - Negative: number analyzed (Participants) | 5 | 6
  Month 12 - Negative | 4 | 2
  Month 12 - Positive Class I: number analyzed (Participants) | 5 | 6
  Month 12 - Positive Class I | 1 | 4
  Month 12 - Positive Class II: number analyzed (Participants) | 5 | 6
  Month 12 - Positive Class II | 0 | 3
  Month 12 - Positive Class I and II: number analyzed (Participants) | 5 | 6
  Month 12 - Positive Class I and II | 0 | 3
  Month 24 - Negative: number analyzed (Participants) | 3 | 3
  Month 24 - Negative | 1 | 1
  Month 24 - Positive Class I: number analyzed (Participants) | 3 | 3
  Month 24 - Positive Class I | 0 | 2
  Month 24 - Positive Class II: number analyzed (Participants) | 3 | 3
  Month 24 - Positive Class II | 2 | 1
  Month 24 - Positive Class I and II: number analyzed (Participants) | 3 | 3
  Month 24 - Positive Class I and II | 0 | 1
  Month 36 - Negative: number analyzed (Participants) | 3 | 3
  Month 36 - Negative | 1 | 1
  Month 36 - Positive Class I: number analyzed (Participants) | 3 | 3
  Month 36 - Positive Class I | 0 | 2
  Month 36 - Positive Class II: number analyzed (Participants) | 3 | 3
  Month 36 - Positive Class II | 2 | 1
  Month 36 - Positive Class I and II: number analyzed (Participants) | 3 | 3
  Month 36 - Positive Class I and II | 0 | 1

5. Secondary Outcome: Number of Infectious Complications
Description: The number of infections complications occurring among study participants is presented here.
Time Frame: Baseline up to Month 36
Measure: Number; unit: complications
Arm/Group | Belatacept Treatment Group | Control Group
Number analyzed (Participants) | 6 | 7
complications | 12 | 18

ADVERSE EVENTS:
Time Frame: Data collection for adverse events began at the Baseline (Day 0) study visit and continued through the Month 36 Study Visit. Data collection for serious adverse events ended 8 weeks after the last administration of the study treatments (up to Month 38).
Description: Adverse events were graded by the physician investigator as follows:
  * Mild (Grade 1): awareness of event but easily tolerated
  * Moderate (Grade 2): discomfort enough to cause some interference with usual activity
  * Severe (Grade 3): inability to carry out usual activity
  * Very Severe (Grade 4): debilitating; significantly incapacitates subject despite symptomatic therapy.
Arm/Group | Belatacept Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 2/6 | 1/7
Serious Adverse Events (participants affected / at risk) | 4/6 | 5/7
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept Treatment Group (N=6) | Control Group (N=7)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 | 0 — secondary to failing graft and end stage renal disease (ESRD)
Groin abscess (Infections and infestations) | 1 | 0
Initiation of hemodialysis (Renal and urinary disorders) | 1 | 0
Deep vein thrombosis and pulmonary embolism (Blood and lymphatic system disorders) | 1 | 0
Peritoneal dialysis catheter blockage or malfunction (Product Issues) | 1 | 1
Exacerbation of hypertension (Vascular disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Acute rejection (General disorders) | 0 | 3
Pericardial effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Peritonitis with sepsis (Infections and infestations) | 0 | 1
Hypertensive crisis with seizure (General disorders) | 0 | 1
Pneumonia related to H1N1 influenza culminating in death (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 — secondary to fatal arrythmia in the setting of ESRD
Infected permacath (Infections and infestations) | 0 | 1
Bacteremia (Infections and infestations) | 1 | 0
Malfunctionig arteriovenous (AV) fistula with edema (Vascular disorders) | 1 | 0
Increased creatinine (Renal and urinary disorders) | 1 | 0
Escherichia coli urinary tract infection (Infections and infestations) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Acute respiratory failure with hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Posterior Reversible Encephalopathy syndrome (General disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept Treatment Group (N=6) | Control Group (N=7)
Pulmonary edema, grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fatigue, grade 1 (General disorders) | 1 | 0
Fatigue, grade 2 (General disorders) | 3 | 0
Nausea, grade 1 (General disorders) | 2 | 2
Abdominal cramps, grade 1 (Gastrointestinal disorders) | 1 | 0
Diarrhea, grade 1 (Gastrointestinal disorders) | 3 | 4
Diarrhea, grade 2 (Gastrointestinal disorders) | 3 | 2
Arthralgia, grade 2 (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia, grade 1 (Musculoskeletal and connective tissue disorders) | 2 | 0
Left leg cramps, grade 2 (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypoglycemia, grade 2 (Metabolism and nutrition disorders) | 2 | 0
Bilateral feet cramps, grade 1 (Musculoskeletal and connective tissue disorders) | 1 | 0
Peritonitis, grade 2 (Infections and infestations) | 3 | 4
Bilateral restless legs, grade 1 (General disorders) | 2 | 0
Forgetfulness, grade 1 (General disorders) | 2 | 0
Disc protrusion, grade 2 (Musculoskeletal and connective tissue disorders) | 1 | 0
Facet joint hypertrophy, grade 2 (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypertension, grade 3 (Vascular disorders) | 1 | 1
Nervousness, grade 1 (General disorders) | 2 | 0
Lesion on upper palate, grade 1 (General disorders) | 1 | 0
Upper respiratory infection, grade 2 (Infections and infestations) | 2 | 0
Upper respiratory infection, grade 1 (Infections and infestations) | 1 | 0
Tendonitis bilateral ankles, grade 1 (Musculoskeletal and connective tissue disorders) | 2 | 0
Chest pain, grade 3 (Cardiac disorders) | 1 | 0
Chest pain, grade 1 (Cardiac disorders) | 1 | 4
Pruritus, grade 2 (Skin and subcutaneous tissue disorders) | 2 | 0
Hypocalcemia, grade 2 (General disorders) | 1 | 0
Abdominal pain, grade 2 (Gastrointestinal disorders) | 1 | 0
Knee meniscus tear, grade 2 (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis in knee, grade 2 (Musculoskeletal and connective tissue disorders) | 1 | 0
Fractured toes due to motor vehicle accident, grade 2 (Injury, poisoning and procedural complications) | 1 | 0
Leg pain possibly due to sciatica, grade 2 (Musculoskeletal and connective tissue disorders) | 2 | 0
Benign right ovarian cysts, grade 1 (Reproductive system and breast disorders) | 1 | 0
Urinary tract infection with bacteremia, grade 3 (Infections and infestations) | 1 | 0
Atrial flutter, grade 1 (Cardiac disorders) | 1 | 0
Squamous cell carcinoma, grades 1 and 2 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anxiety, grade 1 (Psychiatric disorders) | 1 | 0
Peritoneal dialysis site infection, grade 2 (Infections and infestations) | 1 | 0
Coughing and wheezing, grade 2 (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Exacerbation of gout, grades 2 and 3 (Musculoskeletal and connective tissue disorders) | 2 | 0
Multiple non-malignant skin lesions, grade 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Influenza A and B, grade 2 (Infections and infestations) | 1 | 0
Pneumonia, grade 2 (Infections and infestations) | 1 | 0
Burst bursa sac after fall, grade 2 (Injury, poisoning and procedural complications) | 1 | 0
Sycopal episode, grade 3 (General disorders) | 0 | 1
Graft tenderness, grade 1 (General disorders) | 0 | 2
Hematuria, grade 1 (Renal and urinary disorders) | 0 | 2
Posterior reversible encephalopathy, grade 3 (General disorders) | 0 | 1
Peritoneal dialysis catheter malfunction, grade 3 (Product Issues) | 0 | 1
Exacerbation of baseline anemia, grade 2 (General disorders) | 0 | 1
Atrial fibrillation, grade 1 (Cardiac disorders) | 1 | 2
Pericardial effusion, grade 3 (General disorders) | 0 | 1
Shingles, grade 1 (Infections and infestations) | 0 | 2
Pneumonia, grade 3 (Infections and infestations) | 0 | 1
Colitis, grade 3 (Gastrointestinal disorders) | 0 | 1
Cellulitis, grade 2 (Infections and infestations) | 0 | 1
Otitis media, grade 2 (Ear and labyrinth disorders) | 0 | 5
Acute pharyngitis, grade 2 (General disorders) | 0 | 2
Eustacian tube dysfunction, grade 2 (Ear and labyrinth disorders) | 0 | 1
Sinusitis, grade 2 (Infections and infestations) | 0 | 1
Rise in creatinine, grade 2 (Renal and urinary disorders) | 0 | 1
Viral syndrome, grade 2 (Infections and infestations) | 0 | 1
Keratitis dendritic herpes, grade 2 (Eye disorders) | 0 | 1
Hypotension, grade 1 (Vascular disorders) | 0 | 1
Febrile illness, grade 1 (Infections and infestations) | 0 | 2
Shin injury, grade 2 (General disorders) | 0 | 1
Cold sensitivity, grade 1 (General disorders) | 0 | 1
Nausea, grade 3 (General disorders) | 1 | 0
Vomiting, grade 2 (Gastrointestinal disorders) | 1 | 1
Vomiting, grade 3 (Gastrointestinal disorders) | 1 | 0
Diarrhea, grade 3 (Gastrointestinal disorders) | 1 | 0
Lower extremity edema, grade 1 (General disorders) | 4 | 0
Hyperkalemia, grade 2 (General disorders) | 1 | 0
Indigestion, grade 1 (Gastrointestinal disorders) | 1 | 0
Right clogged ear, grade 1 (Ear and labyrinth disorders) | 1 | 0
Hyperphosphatemia, grade 2 (General disorders) | 1 | 0
Hypotension, grade 2 (General disorders) | 1 | 0
Shortness of breath, grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Headache, grade 1 (General disorders) | 1 | 0
Hot flashes, grade 1 (General disorders) | 1 | 0
Intermittent bone pain, grade 1 (Musculoskeletal and connective tissue disorders) | 1 | 0
Intermittent jaw pain, grade 1 (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest wall pain at site of dialysis catheter, grade 1 (Product Issues) | 1 | 0
Scapular pain, grade 1 (Musculoskeletal and connective tissue disorders) | 1 | 0
Chronic pulmonary embolus, grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intermittent hand cramping, grade 1 (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle aches, grade 2 (Musculoskeletal and connective tissue disorders) | 1 | 0
Hyperparathyroidism, grade 2 (Endocrine disorders) | 1 | 0
Asymmetry in right breast, grade 1 (General disorders) | 1 | 0
Hives bilateral lower leg, grade 1 (Skin and subcutaneous tissue disorders) | 1 | 0
Sinus congestion, grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intermittent bilateral foot swelling, grade 1 (General disorders) | 1 | 0
Generalized urticaria, grade 1 (Skin and subcutaneous tissue disorders) | 1 | 0
Lip sore, grade 1 (Skin and subcutaneous tissue disorders) | 1 | 0
Scleral redness, grade 1 (Eye disorders) | 1 | 0
Lower extremity weakness, grade 2 (Musculoskeletal and connective tissue disorders) | 1 | 0
Lower spine pain, grade 2 (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypokalemia, grade 2 (General disorders) | 1 | 0
Urinary tract infection, grade 2 (Infections and infestations) | 1 | 0
Shoulder pain, grade 1 (Musculoskeletal and connective tissue disorders) | 2 | 0
Foot pain, grade 1 (Musculoskeletal and connective tissue disorders) | 1 | 0
Dry cough, grade 1 (General disorders) | 1 | 0
Perihepatic ascites, grade 1 (General disorders) | 1 | 0
Weight loss, grade 2 (General disorders) | 1 | 0
Bilateral hip edema, grade 1 (General disorders) | 1 | 0
Sigmoid diverticulosis, grade 1 (Gastrointestinal disorders) | 1 | 0
Exacerbation of anemia, grade 1 (General disorders) | 1 | 0
Altered mental status, grade 3 (Psychiatric disorders) | 1 | 0
Hypoglycemia, grade 3 (Endocrine disorders) | 1 | 0
Pressure ulcers on sacrum and coccyx, grade 3 (Skin and subcutaneous tissue disorders) | 1 | 0
Weakness, grade 1 (Musculoskeletal and connective tissue disorders) | 1 | 0
Shaking, grade 1 (General disorders) | 1 | 0
Peritoneal catheter removal, grade 1 (General disorders) | 1 | 0
Exacerbation of insomnia, grade 2 (General disorders) | 1 | 0
Weight gain, grade 2 (General disorders) | 1 | 0
Hypertensive crisis, grade 2 (Vascular disorders) | 0 | 2
Hypertension exacerbation, grade 1 (Vascular disorders) | 1 | 0
Syncopal episode, grade 3 (General disorders) | 0 | 1
Fever, grade 2 (General disorders) | 0 | 1
Hypervolemia, grade 1 (General disorders) | 0 | 1
Joint pain, grade 1 (Musculoskeletal and connective tissue disorders) | 0 | 1
Enlarged axillary lymph node, grade 1 (General disorders) | 0 | 1
Pyelonephritis, grade 1 (Renal and urinary disorders) | 0 | 1
Hypokalemia, grade 1 (General disorders) | 0 | 2
Dizziness, grade 1 (General disorders) | 0 | 1
Diaphoresis, grade 1 (General disorders) | 0 | 1
Peritonitis, grade 1 (Infections and infestations) | 0 | 1
Internal hemorrhoids, grade 1 (Gastrointestinal disorders) | 0 | 1
Knee replacement, grade 2 (Surgical and medical procedures) | 0 | 1
Knee drainage, grade 1 (Surgical and medical procedures) | 0 | 1
Lower extremity swelling, grade 1 (General disorders) | 0 | 1
Aortic stenosis, grade 2 (Cardiac disorders) | 0 | 1
Serratia bacteremia, grade 2 (Infections and infestations) | 0 | 1
Metatarsal fracture, grade 2 (Injury, poisoning and procedural complications) | 0 | 1
Lesions removed from arm, grade 2 (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT01921218/Prot_SAP_000.pdf